CLINICAL TRIAL: NCT00429338
Title: Feasibility Study of 3T Endorectal Magnetic Resonance Spectroscopic Imaging (MRSI) of Prostate
Brief Title: 3T Endorectal Magnetic Resonance Spectroscopic Imaging (MRSI) of Prostate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0333
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
Keywords: Genitourinary; Prostate Cancer; Magnetic Resonance Imaging; MRI; Magnetic Resonance Spectroscopic Imaging; MRSI; Endorectal MRSI; Endorectal magnetic resonance spectroscopy imaging; 3 Tesla; 3T Scan; Endorectal coil; Perfluorocarbon compound; PFC; PFC-filled endorectal coil; PFC-MRSI; AIR-MRSI
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR-MRSI (Experimental): Endorectal MRSI with Air
  Interventions: Procedure: AIR-MRSI
- PFC-MRSI (Experimental): Endorectal MRSI with PFC
  Interventions: Procedure: PFC-MRSI

INTERVENTIONS:
Procedure: AIR-MRSI — 3T Magnetic Resonance Spectroscopic Imaging (MSRI) scan performed with an air-filled endorectal coil (AIR-MRSI).
  Other Names: Endorectal magnetic resonance spectroscopy imaging; Magnetic resonance imaging; MRI
  Arms: AIR-MRSI
Procedure: PFC-MRSI — 3T Magnetic Resonance Spectroscopic Imaging (MSRI) scan performed with a perfluorocarbon compound (PFC)-filled endorectal coil (PFC-MRSI).
  Other Names: Endorectal magnetic resonance spectroscopy imaging; Magnetic resonance imaging; MRI
  Arms: PFC-MRSI

SUMMARY:
The objective of this study is to evaluate the feasibility of 3T magnetic resonance spectroscopic imaging (MRSI) of the prostate in improving the spectral resolution, using a perfluorocarbon compound (PFC)-filled endorectal coil.

Specific Aim 1: To compare the spectral quality, measured in Hz (linewidth), of 3T MRSI performed with an air-filled endorectal coil (AIR-MRSI) and a PFC-filled endorectal coil (PFC-MRSI).

Specific Aim 2: To compare the quality of spectra of PFC-MRSI by grading the overall quality of MRSI data of each patient subjectively as being "excellent," "good," "fair," "poor," and "non-diagnostic," based on the status of subjective spectral resolution of Cho, Cr and Po peaks, signal to noise ratio (SNR), baseline distortion, and fat contamination.

DETAILED DESCRIPTION:
MRSI is a type of magnetic resonance imaging (MRI) that uses the same type of scanner as a standard MRI. Unlike standard MRI, which takes pictures of the anatomy (body regions), MRSI takes pictures of the metabolic features of the body. Prostate cancer tissue has certain differences in its metabolism (chemical makeup) that are not seen in normal tissue. MRSI is used to detect prostate tumors by measuring the metabolic features, and an endorectal (inside of the rectum) coil is used. The coil is like an antenna.

Endorectal coils inflated with air are commonly used to detect prostate tumors and measure the status of the disease using a 1.5T (lower-powered, standard clinical) scanner. However, the accuracy of endorectal MRSI scanning still needs improvement. Researchers want to find out if the quality of endorectal MRSI scanning can be improved by using a stronger (3T) scanner and/or using PFC in the endorectal coil instead of air. PFC is a clear and odorless liquid that is known to be virtually non-toxic to the human body. It has been used as an oral contrast (swallowed by mouth) for standard MRIs. As opposed to air, PFC is physically very similar to prostate tissue, which may improve the quality of the MRSI images.

If you agree to take part in this study, you will have 2 endorectal MRSI studies (one with air and one with PFC). The MRSI study with air is diagnostic and considered standard of care, and the MRSI study with PFC is investigational. Before being inserted into your rectum, the coil will be filled with air in order to test for any leakage. You will lie on one side, inside of a 3T MRI scanner, and the coil (covered with protective latex) will be inserted into your rectum. Having the coil inserted is similar to having an enema tip inserted. The coil will be filled with air, and you will lie on your back so the first MRSI study can be completed. The study doctor will carefully check the coil to be sure it is centered at the right place to cover the entire prostate.

After the first MRSI study is completed, the air will be removed using a syringe. The coil will then be filled with PFC, and the second MRSI study will be repeated in the same manner. Once both studies are completed, the coil will be removed after the PFC is removed from the coil. There will be no direct contact between the air or PFC within the coil and your body. In total, the 2 MRSI studies should take about 60 minutes.

After the MRSI studies are completed, researchers will study the information with a special computer to compare the technical quality of the 2 sets of MRSIs. Your participation in this study will be over. Your doctor will receive a report of your diagnostic exam (the MRSI study with air).

This is an investigational study. 3T scanners and the software for routine MRI used for this study are FDA-approved. The use of air in the endorectal coil is a standard procedure. MRSI/MRI equipment for a 1.5T scanner is commercially available and FDA-approved for routine clinical care. PFC used for this study and the software for MRSI acquisition at a 3T scanner have not been FDA-approved. Up to 20 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed biopsy proven prostate carcinoma who are referred to Diagnostic Imaging for magnetic resonance imaging (MRI) / magnetic resonance spectroscopic imaging (MRSI)
2. No previous radiation to prostate or pelvis
3. No hormonal treatment for prostate
4. The interval between the biopsy and magnetic resonance spectroscopic imaging (MRSI): more than 6 weeks
5. Informed consent

Exclusion Criteria:

1. Contraindications for MRI (e.g. cardiac pacemaker)
2. Allergy to Latex
3. Contraindications for magnetic resonance spectroscopic imaging (MRSI) (e.g. history of abdomino-perineal resection of rectum)
4. Metals or any conditions (e.g. hip prosthesis) that can distort the local magnetic field
5. Previous prostate surgery for prostate carcinoma (including, transurethral resection of the prostate (TURP) and cryosurgery), local or systemic treatment for prostate carcinoma (e.g. radiation, androgen deprivation), pelvic radiation (e.g. rectal cancer), rectal surgery, BCG for bladder cancer
6. Children (<18 years)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Spectral quality (linewidth) of 3T MRSI performed with air-filled endorectal coil (AIR-MRSI) and a PFC-filled endorectal coil (PFC-MRSI) | 60 Minutes for 2 sets of MRIs
  Comparison of each linewidths (measured in Hz) between two modalities: endorectal magnetic resonance spectroscopy imaging (MRSI) of prostate using "3 Tesla (3T)" scanner with 1) perfluorocarbon compound (PFC) within endorectal coil versus 2) air.

SECONDARY OUTCOMES:
Total number of patients for each grade from each group with AIR-MRSI and PFC-MRSI | Patients: 60 Minutes for 2 sets of MRIs; Study Duration 4 Years
  The quality of PFC-MRSI and AIR-MRSI will be graded subjectively as being "excellent," "good," "fair," "poor," and "non-diagnostic," based on the status of subjective spectral resolution of Cho, Cr, Po, and Ci peaks, signal-noise-ratio (SNR), baseline distortion, and fat and seminal vesicle contaminations.

CONTACTS AND LOCATIONS:
Overall Officials: Haesun Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org